CLINICAL TRIAL: NCT02545686
Title: Use of the Real-time Position Management (RPM) to Measure the Effects of Continuous Positive Airway Pressure (CPAP) on Duration of Breath Hold and Diaphragm Motion in Normal Volunteers
Brief Title: Effect of CPAP on Breath Hold and Chest Movement in Normal Volunteers
Acronym: CPAP_normal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SHEBA-15-2364-YL-CTIL
Record Dates: First submitted 2015-09-02; First posted 2015-09-10 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteers; Effect of CPAP on Chest Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one (Experimental): this is a single arm study. All subjects treated the same way, and undergo four interventions:
  1. Chest wall movement assessment without CPAP
  2. Breath hold assessment without CPAP
  3. Chest wall movement assessment with CPAP
  4. Breath hold assessment with CPAP
  Interventions: Behavioral: Chest wall movement assessment without CPAP; Behavioral: Breath hold assessment without CPAP; Procedure: Chest wall movement assessment with CPAP; Procedure: Breath hold assessment with CPAP

INTERVENTIONS:
Behavioral: Chest wall movement assessment without CPAP — While subject is breathing normally, determine chest wall movement (via RPM waveform) with free breathing, over the course of half an hour.
Behavioral: Breath hold assessment without CPAP — While subject is breathing normally, subject will perform a moderate and a deep inspiratory breath hold. Duration, reproducibility and tolerance of deep inspiratory breath hold will be recorded.
Procedure: Chest wall movement assessment with CPAP — While subject is breathing via CPAP machine, determine chest wall movement (via RPM waveform) with free breathing, over the course of half an hour.
Procedure: Breath hold assessment with CPAP — While subject is breathing via CPAP machine, subject will perform a moderate and a deep inspiratory breath hold. Duration, reproducibility and tolerance of deep inspiratory breath hold will be recorded.

SUMMARY:
CPAP will be applied to normal volunteers inorder to understand CPAP's effects on breathing and chest wall motion.

DETAILED DESCRIPTION:
CPAP is a non-invasive ventilation technique that is commonly used to treat sleep apnea. Using a small air-pump, tubing and facemask, it provides a constant stream of pressurized air to the upper airways and lungs. Some of the physiological effects noted during CPAP are hyperinflation of the lungs, stabilizing and flattening of the diaphragm, and decrease in tidal volume. The effects on duration of breath hold are unknown. During radiation treatment, these effects are expected to reduce tumor and organ motion which reduces the volume of normal tissue being irradiated and also creates favorable treatment geometry by moving the heart away from the anterior chest wall. An important advantage of CPAP compared to other techniques is that active patient cooperation is not required. The potential exists to combine use of CPAP with other respiratory management techniques such as breath hold and improve overall effectiveness. When used in sleep apnea it is well tolerated and poses little risk to patients. There are no published reports of the use of CPAP in radiation therapy.

In initial studies the Varian RPM system was used to assess respiratory motion with and without CPAP for patients receiving radiation therapy. This commercially available, non-invasive system works by directing an infrared beam onto an infrared motion detector that is placed on the patients' upper abdomen. The detector records the change in abdomen position that occurs with respiration as a change in amplitude of the detector position. Interventions that effect respiration will be recorded by an increase or decrease in the amplitude of the detector motion. When used in breath hold, the detector remains in a fixed position with a very narrow gating window.

Based on initial experience with the RPM system, it has been found that approximately 1 hour of CPAP use is required to reduce diaphragm motion. Although early results are favorable using this approach, it is not certain that this is the best or most efficient method of use for all patients. The use of CPAP combined with breath hold techniques has not been studied.

The objectives of this study are to use the RPM system in normal volunteers to:

1. Study the effects of CPAP on diaphragm motion to allow better optimization for the use of CPAP as a respiratory management technique during free breathing.
2. Determine the feasibility of use of CPAP as a respiratory aid for use in patients treated with breath hold techniques. Determine the effects of CPAP on duration; reproducibility and tolerance of the breath hold technique.

ELIGIBILITY:
Inclusion Criteria:

* Normal volunteers without a cancer diagnosis.
* No contraindications to the use of CPAP

  * Facial injury or deformity preventing wearing facial mask
  * Recurrent vomiting
  * Chronic cough with phlegm
  * Previous pneumothorax
  * Facial lacerations or fractures
  * Recent tracheal or esophageal anastomosis
  * Recent GI surgery (last 90 days).
* 18-90 years of age
* Ability to sign informed consent
* Hebrew or English speakers

Exclusion Criteria:

* Contraindications to CPAP

  * Facial injury or deformity preventing wearing facial mask
  * Recurrent vomiting
  * Chronic cough with phlegm
  * Previous pneumothorax
  * Facial lacerations or fractures
  * Recent tracheal or esophageal anastomosis
  * Recent GI surgery (last 90 days).
* Under age 18 or above age 90 years
* Inability to sign informed consent
* Members of special populations (mental illness, pregnant women, prisoners, not legally competent).
* History of severe active restrictive or obstructive lung disease (as defined as at least one hospitalization over previous two years)
* Any medical condition requiring an inpatient hospitalization for more than 72 hours over the previous 2 years, aside from elective surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Chest wall motion amplitude | 2 hours
  Amplitude of chest wall motion, measured in centimeters.

SECONDARY OUTCOMES:
Duration of breath hold | 2 hours
  Length (in seconds) that are subjects able to hold their breath.
Reproducibility of breath hold depth | 2 hours
  When 'breath hold' is performed three consecutive times, ascertain if it performed to the same depth each time. Measured in centimeters.
Respiratory rate | 2 hours
  Number of breaths per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Goldstein, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel